CLINICAL TRIAL: NCT03133208
Title: Serum Biomarkers in Sepsis Associated Encephalopathy (SAE)
Brief Title: Sepsis Associated Encephalopathy (SAE) Biomarkers
Status: Active, not recruiting | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201700135
Record Dates: First submitted 2017-04-10; First posted 2017-04-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Sepsis; Altered Mental Status; Sepsis-Associated Delirium; Sepsis Associated Encephalopathy; Delirium, Sepsis Associated
Keywords: sepsis; sepsis associated encephalopathy; sepsis associated delirium; altered mental status
MeSH Terms: conditions — Sepsis; Sepsis-Associated Encephalopathy | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples (serum).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sepsis with AMS: Patients presenting to the ED with suspected sepsis who develop altered mental status
  Interventions: Procedure: Blood draws
- Sepsis without AMS: Patients presenting to the ED with suspected sepsis without change in mental status
  Interventions: Procedure: Blood draws
- Control: Patients presenting to the ED with no suspicion of systemic inflammation that need hospitalization (control category)
  Interventions: Procedure: Blood draws

INTERVENTIONS:
Procedure: Blood draws — Blood draws will be collected via venipuncture or IV at hours 0, 6, 12, 18, 24, 48, 72 (7 draws total). Each draw would be up to 20 mL of blood (but no less than 10 mL).

SUMMARY:
Sepsis associated encephalopathy (SAE) is a poorly understood acute cerebral dysfunction that frequently appears in the setting of sepsis induced systemic inflammation. In fact, altered mentation is recognized as an independent predictor of death and poor outcomes in patients with sepsis. SAE may be manifested by a number of symptoms characterized by a change in baseline behavior, attention, alertness, cognition, or executive functioning. It occurs in the absence of direct Central Nervous System (CNS) infection, and the exact pathophysiology is of SAE is unknown, but theoretically seems to encompass a constellation of mechanisms such as impairment of the blood brain barrier (BBB), endothelial dysfunction, alteration in cerebral blood flow and neurotransmission, circulating inflammatory mediators, cellular hypoxia, and metabolic disturbances, that ultimately result in neuronal dysfunction and cell death. SAE is characterized by an altered mental status (AMS) that ranges from delirium to coma, and can lead to long-term cognitive impairment. SAE may appear early in the course of sepsis, and is often underestimated as an independent factor of mortality, yet the pathophysiology of SAE remains unknown, and there is a lack of specific investigations available to clinicians. Studies have evaluated biomarkers as prognostic tools. The Investigator propose to measure neuron specific enolase (NSE), S-100B, glial fibrillary acidic protein (GFAP), ubiquitin C-terminal hydrolase L1 (UCH-L1), Tau protein, Copeptin, spectrin breakdown products (SBDP 145, SBDP150), αII-spectrin N-terminal fragment (SNTF), neurofilament light and heavy chains (NF-L, NF-H), myelin basic protein (MBP), secretoneurin (SN), and other peptide levels in the serum of sepsis patients who develop altered mental status, to evaluate the kinetics of said biomarkers for 72 hours. The Investigator will monitor the course of the patients' hospitalization to determine whether there are biomarker correlates with survival and outcomes, including neurologic impairment. Finally, this investigation may provide a mechanistic pathway that defines the development of AMS in septic patients.

DETAILED DESCRIPTION:
Sepsis associated encephalopathy (SAE) is a common neurological complication of sepsis that is often associated with worse prognosis, yet remains poorly understood. It occurs in the absence of direct brain infection or other types of disease-associated encephalopathy such as hepatic or renal encephalopathy, and is a result of systemic inflammation (1). Clinically, a diagnosis of SAE is made when there is an impaired mental state in the presence of an extracranial infection. Clinical features of SAE include change in mental status (altered mental status/ AMS), disturbances in mental processes, agitation, disorientation, impaired attention, hypersomnolence, delirium or coma. SAE may be an early sign of sepsis that is manifested prior to overt evidence of other organ failures (2), and is an independent prognosticator of morbidity and mortality (3). Moreover, sepsis survivors can suffer from long-term cognitive impairments that impact their quality of life.

The pathophysiology of SAE is a complex constellation of proposed mechanisms that include direct insult to brain tissue from circulating inflammatory mediators that are overexpressed in sepsis, disturbances in metabolic pathways, cellular hypoxia, disruption of the BBB integrity, alterations in neurotransmission, impairment of regulation of the brain perfusion. The consequence of this combination of neuroinflammatory and ischemic processes is neuronal degeneration and cell death (apoptosis).

It is difficult to diagnose SAE early, as sepsis is often a diagnosis of exclusion and can be occult in presentation. For example, emergency physicians may conduct diagnostic studies to evaluate for stroke, metabolic disturbance (i.e. hyponatremia, hypoglycemia, vitamin deficiency, medication reaction), toxicity, seizure or other acute neurologic condition. In addition, severe sepsis patients may be intubated and are often sedated, which poses a challenge to conducting a neurological assessment of their mental status. There may be changes in electroencephalography (EEG), somatosensory-evoked potentials (SSEP), or neuroimaging but these tests lack specificity and SAE remains a diagnosis of exclusion.

Injured neurons release neuron specific proteins that diffuse across the disrupted BBB into the blood and could have diagnostic relevance in diagnosing SAE. Neuron specific enolase (NSE) and S100 beta (S100B) are biomarkers currently used in the setting of SAE and have been studied clinically. There is a lack of human studies on other proteins such as GFAP, co-peptin, Tau, neurofilament light/ heavy chain, UCH-L1, SBDP, MBP, and secretoneurin that have been proposed as potential biomarkers of neurological outcome for other causes of acute brain dysfunction such as traumatic brain injury (TBI) and hypoxic ischemic encephalopathies (HIE) and could potentially serve as candidate biomarkers to diagnose SAE.

Most studies lack a control cohort. The Investigator intends to sample sepsis patients that present to the emergency department but do not develop altered mental status within our study as well.

The Investigator therefore propose a prospective, observational study in which the study team will perform blood biomarker analysis from time of enrollment up to study day 3. This would be done by drawing blood at (0-30mins), and additional blood draws at hours 6, 12, 18, 24, 48, 72. The Investigator will then determine whether biomarker levels correlate with neurologic assessment in the Emergency Department (ED), degree of overall organ dysfunction, survival to hospital admission, survival to hospital discharge, and functional neurologic outcome at discharge and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

* ≥ 18 years old
* Presented to the emergency department at Shands
* Has not donated blood within the last 8 weeks
* Willing to participate and follow up at 6 months after discharge from the hospital
* Not anemic or have any other hematological disorders that requires transfusions

Meets two or more Systemic Inflammatory Response Syndrome (SIRS) criteria:

* Temperature >38°C or <36°C
* Heart rate (HR) > 90bpm
* Respiratory rate (RR) > 20bpm or partial pressures of carbon dioxide (PaCO2) <32mm mercury (HG)
* White Blood Cell (WBC) >12,000/µL or < 4,000/µL or >10% immature/ bands Clinical suspicion of sepsis (blood cultures ordered/ antibiotics started) Altered mental status Enrolled within 6 hours of ED presentation

Cohort 2

* ≥ 18 years old
* Presented to the emergency department at Shands
* Has not donated blood within the last 8 weeks
* Willing to participate and follow up at 6 months after discharge from the hospital
* Not anemic or have any other hematological disorders that requires transfusions

Meets two or more SIRS criteria:

* Temperature >38°C or <36°C
* HR > 90bpm
* RR > 20bpm or PaCO 2 <32mmHG
* WBC >12,000/µL or < 4,000/µL or >10% immature/ bands Clinical suspicion of sepsis (blood cultures ordered/ antibiotics started) No altered mental status Enrolled within 6 hours of ED presentation

Cohort 3 (control)

* Does not meet SIRS criteria
* No clinical suspicion of sepsis (no cultures/ antibiotics ordered)
* Not altered
* Patient has admission orders

Exclusion Criteria (all cohorts):

* Participating in another interventional, therapeutic study that may affect the results of this study
* Subject has neurodegenerative disease or other neurological disorder (dementia, Parkinson's disease, multiple sclerosis, seizure disorder, or brain tumours)
* History of neurosurgery within the last 30 days
* Acute brain injury within the last 30 days (ischemic/ haemorrhagic stroke, traumatic brain injury)
* Subject is anemic OR donated blood within the last 8 weeks OR has a hematological disorder that requires transfusions
* Subject has history of liver failure OR renal failure
* Pregnant or lactating female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to UF Health Shands emergency department with sepsis. The sepsis cohort will be further broken down into sub- cohorts:
  * Cohort 1: Patients who present with altered mental status
  * Cohort 2: Patients who do not present with altered mental status A control cohort (cohort 3) will include patients presenting to the ED with no suspicion of systemic inflammation that need hospitalization.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Relationship between biomarkers and neurological outcome- Delirium | 1 year
  Acute encephalopathy will be measured using the mental status assessment including the Delirium Triage Screen (DTS) Brief Confusion Assessment Method (bCAM). DTS-bCAM assessment is a flowchart that helps diagnose a patient who is altered.
Relationship between biomarkers and neurological outcome - Blessed | 1 year
  Acute encephalopathy will be measured using the mental status assessment short blessed test (SBT). Sum Total (range 0-28) [0-4 = normal cognition, 5-9 = questionable impairment, ≥ 10 = Impairment consistent with dementia]

SECONDARY OUTCOMES:
Relationship between biomarkers and organ dysfunction | 1 year
  Organ dysfunction will be assessed using Sequential Organ Failure Assessment (SOFA) methodology, a mortality assessment tool that monitors the dynamics of cardiovascular, respiratory, neurological, renal, hepatic, and hematological organ function.
Relationship between biomarkers and overall survival | 7-day, 28-day, and 6-months mortality
  Date of death will be recorded for all patients who died during the study period. Rate of survival will be assessed.
Degree of neurological impairment | up to 2 weeks
  assessed using the Cerebral Performance Category (CPC) scoring [CPC 1: A return to normal cerebral function and normal living, CPC 2: Cerebral disability but sufficient function for independent activities of daily living, CPC 3: Severe disability, limited cognition, inability to carry out independent existence, CPC 4: Coma, CPC 5: Brain death
Degree of neurological impairment | 6 months after discharge
  Cognitive Failure Questionnaire (CFQ) sum of 25 questions, range 0-100 assessing Forgetfulness, Distractibility, and False Triggering

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Carmelle Elie, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chaudhry N, Duggal AK. Sepsis Associated Encephalopathy. Adv Med. 2014;2014:762320. doi: 10.1155/2014/762320. Epub 2014 Sep 30. PMID 26556425
- [Background] Bello JH, Park M. Sepsis-associated encephalopathy as a differential diagnosis with motor deficit plus altered mental status. Clinics (Sao Paulo). 2007 Apr;62(2):199-202. doi: 10.1590/s1807-59322007000200017. No abstract available. PMID 17505707
- [Background] Sprung CL, Peduzzi PN, Shatney CH, Schein RM, Wilson MF, Sheagren JN, Hinshaw LB. Impact of encephalopathy on mortality in the sepsis syndrome. The Veterans Administration Systemic Sepsis Cooperative Study Group. Crit Care Med. 1990 Aug;18(8):801-6. doi: 10.1097/00003246-199008000-00001. PMID 2379391
- [Background] Shankar-Hari M, Rubenfeld GD. Understanding Long-Term Outcomes Following Sepsis: Implications and Challenges. Curr Infect Dis Rep. 2016 Nov;18(11):37. doi: 10.1007/s11908-016-0544-7. PMID 27709504
- [Background] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258
- [Background] Papadopoulos MC, Davies DC, Moss RF, Tighe D, Bennett ED. Pathophysiology of septic encephalopathy: a review. Crit Care Med. 2000 Aug;28(8):3019-24. doi: 10.1097/00003246-200008000-00057. PMID 10966289
- [Background] Consales G, De Gaudio AR. Sepsis associated encephalopathy. Minerva Anestesiol. 2005 Jan-Feb;71(1-2):39-52. English, Italian. PMID 15711505
- [Background] Jacob A, Brorson JR, Alexander JJ. Septic encephalopathy: inflammation in man and mouse. Neurochem Int. 2011 Mar;58(4):472-6. doi: 10.1016/j.neuint.2011.01.004. Epub 2011 Jan 8. PMID 21219956
- [Background] Davies DC. Blood-brain barrier breakdown in septic encephalopathy and brain tumours. J Anat. 2002 Jun;200(6):639-46. doi: 10.1046/j.1469-7580.2002.00065.x. PMID 12162731
- [Background] Polito A, Eischwald F, Maho AL, Polito A, Azabou E, Annane D, Chretien F, Stevens RD, Carlier R, Sharshar T. Pattern of brain injury in the acute setting of human septic shock. Crit Care. 2013 Sep 18;17(5):R204. doi: 10.1186/cc12899. PMID 24047502
- [Background] Zhang QH, Sheng ZY, Yao YM. Septic encephalopathy: when cytokines interact with acetylcholine in the brain. Mil Med Res. 2014 Sep 1;1:20. doi: 10.1186/2054-9369-1-20. eCollection 2014. PMID 25722876
- [Background] Szatmari S, Vegh T, Csomos A, Hallay J, Takacs I, Molnar C, Fulesdi B. Impaired cerebrovascular reactivity in sepsis-associated encephalopathy studied by acetazolamide test. Crit Care. 2010;14(2):R50. doi: 10.1186/cc8939. Epub 2010 Mar 31. PMID 20356365
- [Background] Sharshar T, Annane D, de la Grandmaison GL, Brouland JP, Hopkinson NS, Francoise G. The neuropathology of septic shock. Brain Pathol. 2004 Jan;14(1):21-33. doi: 10.1111/j.1750-3639.2004.tb00494.x. PMID 14997934
- [Background] Bozza FA, D'Avila JC, Ritter C, Sonneville R, Sharshar T, Dal-Pizzol F. Bioenergetics, mitochondrial dysfunction, and oxidative stress in the pathophysiology of septic encephalopathy. Shock. 2013 May;39 Suppl 1:10-6. doi: 10.1097/SHK.0b013e31828fade1. PMID 23481496
- [Background] Hirota K. Involvement of hypoxia-inducible factors in the dysregulation of oxygen homeostasis in sepsis. Cardiovasc Hematol Disord Drug Targets. 2015;15(1):29-40. doi: 10.2174/1871529x15666150108115553. PMID 25567333
- [Background] Shehabi Y, Riker RR, Bokesch PM, Wisemandle W, Shintani A, Ely EW; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Delirium duration and mortality in lightly sedated, mechanically ventilated intensive care patients. Crit Care Med. 2010 Dec;38(12):2311-8. doi: 10.1097/CCM.0b013e3181f85759. PMID 20838332
- [Background] Iacobone E, Bailly-Salin J, Polito A, Friedman D, Stevens RD, Sharshar T. Sepsis-associated encephalopathy and its differential diagnosis. Crit Care Med. 2009 Oct;37(10 Suppl):S331-6. doi: 10.1097/CCM.0b013e3181b6ed58. PMID 20046118
- [Background] Sonneville R, Verdonk F, Rauturier C, Klein IF, Wolff M, Annane D, Chretien F, Sharshar T. Understanding brain dysfunction in sepsis. Ann Intensive Care. 2013 May 29;3(1):15. doi: 10.1186/2110-5820-3-15. PMID 23718252
- [Background] Bone RC, Balk RA, Cerra FB, Dellinger RP, Fein AM, Knaus WA, Schein RM, Sibbald WJ. Definitions for sepsis and organ failure and guidelines for the use of innovative therapies in sepsis. The ACCP/SCCM Consensus Conference Committee. American College of Chest Physicians/Society of Critical Care Medicine. Chest. 1992 Jun;101(6):1644-55. doi: 10.1378/chest.101.6.1644. PMID 1303622
- [Background] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL; International Surviving Sepsis Campaign Guidelines Committee; American Association of Critical-Care Nurses; American College of Chest Physicians; American College of Emergency Physicians; Canadian Critical Care Society; European Society of Clinical Microbiology and Infectious Diseases; European Society of Intensive Care Medicine; European Respiratory Society; International Sepsis Forum; Japanese Association for Acute Medicine; Japanese Society of Intensive Care Medicine; Society of Critical Care Medicine; Society of Hospital Medicine; Surgical Infection Society; World Federation of Societies of Intensive and Critical Care Medicine. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Crit Care Med. 2008 Jan;36(1):296-327. doi: 10.1097/01.CCM.0000298158.12101.41. PMID 18158437